CLINICAL TRIAL: NCT02518074
Title: Hearing and Vestibular Interactions in the Collection of Own Body and Sense of Self
Acronym: AUDIOSELF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-070
Record Dates: First submitted 2015-07-22; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Hearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HEARING AND VESTIBULAR INTERACTIONS (Other): Hearing and Vestibular Interactions during two body positions (standing / supine) and three gravity conditions (weightlessness hyper gravity and normal gravity).
  Interventions: Other: Hearing and Vestibular Interactions

INTERVENTIONS:
Other: Hearing and Vestibular Interactions — in two body positions (standing / supine) and three gravity conditions (weightlessness hyper gravity and normal gravity).
  Other Names: in two body positions and three gravity conditions

SUMMARY:
The investigators objective is twofold. Investigators propose to study how the vestibular and auditory information interact in the construction of coherence between the staff and extrapersonal space.

Furthermore, investigators want to investigate whether, even in the absence of gravity, the auditory spatial information allocentric provide a framework for spatial reference.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged between 18-65 years
* Affiliates to a social security system or, for non-residents in France, holder of a European Health Insurance Card European (EHIC European Health Insurance Card)
* Who are willing to take part in the study,
* Who gave written informed consent,
* Declared fit after a similar visit to a medical aeronautical medical fitness for the non-professional cabin crew in civil aviation. There will be no other aptitude tests for the selection of subjects.

Exclusion Criteria:

* People who took part in a biomedical research protocol for which the exclusion period is complete,
* People with psychotic disorders and / or depression,
* People receiving psychotropic medication,
* People with alcohol dependence or illicit substances,
* People with visual acuity less than 8 / 10ths corrected by lenses or glasses,
* People with a significant decrease in hearing,
* pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Responses to the questionnaire "Botvinick Cohen" on the sensations of the body out experiments | baseline
Answers on the location of auditory stimuli | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France